CLINICAL TRIAL: NCT05809258
Title: Comparison of Efficacy of Ultrasound-Guided Supraclavicular and Axillary Block for Arterio-Venous Fistula Creation: An Observer-Blinded, Non-inferiority Randomized Controlled Trial
Brief Title: Supraclavicular Versus Axillary Block for Arteriovenous (AV) Fistula Creation
Acronym: CUGSCAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr Jyoti Burad, Senior specialist, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 061/2023
Record Dates: First submitted 2023-02-22; First posted 2023-04-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Arteriovenous Fistula; Brachial Plexus Block; Clinical Efficacy
Keywords: Arteriovenous fistula; brachial plexus block; ultrasound guided; complications; block recovery
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Brachial Plexus Block

STUDY DESIGN:
Intervention Model Description: Two parallel arms of interventions, no crossover.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and assessor will be blinded. The block performer anaesthetist and the patient will know the technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraclavicular block (Active Comparator): In the supraclavicular group, the ultrasound probe will be positioned in the supraclavicular fossa, pointing caudad and locating the subclavian artery. The first rib is identified deep to the artery, and the hyperechoic pleura will be identified by sliding lung sign. The brachial plexus is consistently found with a characteristic ''honeycomb'' appearance lateral and superficial to the subclavian artery and superior to the first rib. The needle will be introduced through the skin from lateral to medial, in-plane with the transducer, with constant visualization, and directed toward the deep border of the nerve group. Three separate injections will be made at various sites in the bundle, tending to start deep, in the ''corner pocket'' close to the artery, and moving more superficially. The local anesthetics will be Lidocaine 2% 10 ml + Levobupivacaine 0.5% 10 ml.
  Interventions: Procedure: Supraclavicular block
- Axillary block (Active Comparator): Patients in the axillary group are placed in the supine position with the arm to be blocked, abducted and externally rotated. After sterilization of the axilla, the Ultrasound probe will be placed parallel to the anterior axillary fold at the axilla to identify the axillary artery and surrounding radial, ulnar, and median nerve, appearing as hypo-echoic round structures around the axillary artery. The musculocutaneous nerve will also be identified between the coracobrachialis and biceps muscle or in either of them. Lidocaine 1% was infiltrated subcutaneously 1 cm lateral to the probe, and then 0.5% bupivacaine will be injected around branches of the brachial plexus. The local anesthetics will be Lidocaine 2% 10 ml + Levobupivacaine 0.5% 15 ml. In this block, 5-7 ml of local anesthetic will block each nerve.
  Interventions: Procedure: Axillary block

INTERVENTIONS:
Procedure: Supraclavicular block — brachial plexus nerve block by supraclavicular route
  Other Names: brachial plexus block
  Arms: Supraclavicular block
Procedure: Axillary block — brachial plexus nerve block by axillary route
  Other Names: brachial plexus block
  Arms: Axillary block

SUMMARY:
This study compares the analgesic efficacy of supraclavicular brachial plexus nerve block to axillary nerve block techniques in adults undergoing AV fistula creation. Both these techniques will be done under ultrasound guidance, using the same local anesthetic drug. 120 patients will be included in this study, 60 patients for each technique. This study will help us know better regional anesthesia techniques, the additional need for analgesia/anesthesia, and the recovery rate following either of the blocks for AV fistula surgery. An interim analysis will be done after recruiting 50% of cases (30 cases) in both arms.

DETAILED DESCRIPTION:
Introduction An AV fistula creation is generally performed at the antecubital fossa under regional anesthesia. General anesthesia is associated with increased cardiorespiratory complications in patients with end-stage renal disease. Thus, in such patients, RA, such as a brachial plexus block (BPB), is favored for AVF creation. In this study comparison between two well-established and frequently used approaches of brachial plexus block: supraclavicular and axillary, will be compared.

The supraclavicular block is one of several approaches used for the brachial plexus block. The block is performed at the level of the brachial plexus trunks, where almost the entire sensory, motor, and sympathetic innervation of the upper extremity is carried in just three nerve structures confined to a very small surface area. Indications for the supraclavicular block include elbow, forearm, and hand surgeries.

The axillary block technique is relatively easy to approach and simple to perform and may be associated with a lower risk of complications than supraclavicular BPB. The supraclavicular has a slightly wider area of coverage and a supposedly higher rate of complications compared to the axillary approach when performed with a traditional approach without ultrasound guidance. Using ultrasound should reduce the rate of complications for both blocks. No randomized control study has compared the efficacy of both blocks for AV Fistula creation with ultrasound guidance. This study aims to determine a better anesthesia technique for AV fistula creation in terms of anesthesia efficacy, complications, and recovery.

Method

Study type: Randomized, Controlled, observer-blinded non-inferiority trial, with two parallel arms.

Blinding: The observer, Anesthetist 2, and data analyst will be blinded. But the patient and the block performer both will know the block group.

Randomization: The statistician will generate the block randomization sequence, and the file will be handed over to the principal investigator. The file will be accessed during randomization, and group allocation will be obtained and conveyed to the block performer (Anesthetist 1). The remaining will be kept securely with the principal investigator. The patient will be randomized into groups A (supraclavicular nerve block) and B (axillary nerve block). The randomization sequence will be kept locked with a password-protected file.

Crossover: Nil Study duration: Prospective for 18-24 months, depending on the case recruitment rate.

Number of groups: 2 Sample size: 120 cases, 60 in each group. Assessment: The patient will be assessed intraoperatively at 10 minutes after the block and every 5 minutes. The final assessment of block adequacy will be done 30 minutes after the block, and a decision will be taken on adequacy. The next assessment will be at two hours and 30 minutes after time 0 and will continue every hour till complete recovery of the block in PACU and ward.

Target follow-up duration: The patient will be followed till complete recovery of muscle power of the upper limb.

Eligibility Study Population: all adult>18 years old patients posted for AV fistula creation in the antecubital fossa.

Inclusion Criteria:

* Age >18 years old
* Patients undergoing AV fistula creation in the antecubital fossa

Exclusion Criteria:

* Patient Refusal
* Hemodynamically unstable patient
* Local infection over the insertion site
* Coagulopathy
* Known allergy to Local Anaesthetic medications.
* Grossly abnormal anatomy
* Severe chronic airways disease

Primary Outcome:

• Requirement of additional analgesics intraoperatively or block failure (conversion to general anesthesia)

Secondary outcome:

* Time of motor recovery of block
* Rate of complications
* Comparison of change in brachial artery diameter at the elbow before and after block

Study population:

Sample size The estimated sample size is 120 (60 in each group). The estimation was based on the success rate reported in the literature (95%), the non-inferiority margin between supraclavicular and axillary brachial plexus block to be < 10%. The power was set at 80%, and the alpha error was set at 5%. The allocation ratio was 1:1. The software used for the sample size calculation is nMaster 2.0 sample size calculator.

Method:

Patients will be posted for surgery in the operating room list. An appropriate population, as per eligibility criteria, will be approached. An explanation of the study will be done in comprehensive language. The patient's rights will be explained to the patient/relatives. Informed consent will be taken on the consent form. As per the departmental schedule and protocol, a separate anesthetist will do the pre-anesthetic checkups. On the day of surgery, the patient will be premedicated per standard institutional guidelines; the intravenous cannula will be inserted in the ward. On arrival of the patients to the operative theatre, ASA monitors will be attached (ECG, non-invasive blood pressure, and SpO2). The patient will be positioned for the block, and the largest brachial artery diameter will be recorded with the help of the ultrasound. This will be done before attempting block, at the start and end of surgery. Following the study protocol, the block will be given as per randomization by one of the expert anesthesia consultants (Anesthetist 1). The supraclavicular and axillary block sites will be dressed for all patients to avoid disclosing the technique to Anesthetist 2 and the assessors. An independent observer will record all the timings and procedure details. At the end of the procedure, the patient will be shifted to PACU (Post-Anesthesia Care Unit).

Assessment of the block: The block assessment will start after 10 minutes of finishing the block (Time 0) and will be repeated every 5 minutes until the start of surgery. If the anesthesia state is not achieved within 30 minutes of the block, rescue analgesia or general anesthesia will be given. Rescue analgesia will be given when the block is incomplete (only one segment/nerve dermatome will be spared). It will consist of Fentanyl 0.5 mics/kg aliquots followed by local infiltration with 1% Lidocaine by the surgeon and Paracetamol 15 mg/kg in the same sequence, one after another if previous rescue analgesia is not effective. General anesthesia will be given if there is a complete block failure (defined as no block in more than one nerve).

Assessment of the block intraoperatively: The muscle power will be checked by asking the patient to flex and extend his forearm and adduct, abduct and oppose the thumb and all fingers. Motor blockade of the musculocutaneous nerve will be checked by elbow flexion, ulnar nerve by thumb adduction, radial by thumb abduction and median nerve by thumb opposition. The power will be graded on a three-point scale: 0=no block, 1=paresis, and 2=paralysis. Whereas sensory blockade will be assessed on another three-point scale with a cold test: 0=no block, 1=analgesia (can feel touch but not cold), and 2=anesthesia (cannot feel touch).

Assessment of the block postoperatively: The assessment will start two hours 30 minutes after time 0 and will continue every hour till discharge or complete recovery of the block.

Possible Complications:

* Pneumothorax
* Horner syndrome
* Vascular puncture and Hematoma
* Diaphragmatic paralysis
* Local anesthetic systematic toxicity (LAST)
* Prolonged block recovery

Troubleshooting:

Pneumothorax: Because of the proximity of the pleura to the brachial plexus at the clavicle's level, the lung's apex can be damaged. It is a rare complication; pneumothorax was a more frequent complication of the supraclavicular block before ultrasound use, with a reported incidence of 0.6% to 6.1%. Maintaining needle tip visibility at all times during needle advancement is critical while performing US-guided block., An urgent chest radiograph (CXR) will be requested if the pleura is punctured, and supplemental oxygen will be delivered. A general surgeon will insert a chest tube under local anaesthesia and connect to suction at a negative pressure of 20 cm H2O. A repeat CXR will be done to confirm the correct position of the chest tube and re-expansion of the lung. The chest tube will be removed a few days later upon the resolution of symptoms.

Horner's syndrome may correspond to the diffusion of local anaesthetics in prevertebral spaces, ultimately involving the sympathetic nerves and communicating with cervical nerve trunks. It results from paralysis of the ipsilateral sympathetic cervical chain (stellate ganglion) caused by surgery, drugs (mainly high concentrations of local anaesthetics), local compression (hematoma or tumour), or inadequate perioperative positioning of the patient. It appears after the block with a specific triad (ptosis, miosis, and exophthalmos) and quickly disappears without any sequelae. Horner's syndrome may be described as an unpleasant side effect because it has no clinical consequences, and if it occurs, patients should be reassured and monitored closely.

Vascular puncture and Hematoma: These are not commonly encountered with ultrasound guidance. Bleeding can be controlled by pressure, conservative treatment and surgical exploration if needed. Especially if a hematoma forms, it should be removed promptly. Comprehensive knowledge of anatomy and skills is crucial to avoid nerve injuries, so the blocks will be performed by experts and US-guided in this study.

Diaphragmatic paralysis: the phrenic nerve lies in front of the anterior scalene muscle, and local anaesthetic injected around the proximal, i.e., interscalene, part of the plexus can, therefore, easily affect the phrenic nerve. Treatment is conservative and usually resolves within a few days to weeks. Ultrasonography was chosen to demonstrate diaphragmatic movement as it reliably shows the paradoxical movement of the diaphragm in the event of paralysis.

LAST: It is rare as the blocks are usually US-guided, and drugs are given in smaller amounts than the toxic levels and given with frequent aspirations to prevent injecting into blood vessels.

The following actions will be taken when managing local anaesthetic toxicity:

* Stop the local anaesthetic injection.
* Institute basic life support and call for assistance.
* Secure the airway, ventilate with 100% oxygen, and gain intravenous access.
* Seizures can be managed with a benzodiazepine or anaesthetic induction agent.
* If a cardiac arrest has occurred, commence advanced life support.
* Note that arrhythmias are often refractory, and resuscitation should be prolonged.
* Treatment with IntraLipid: An initial dose of 20% lipid emulsion at 1.5 ml/kg or a 100 ml bolus can be administered over a few minutes. This can be repeated after 5 minutes two or more times for persistent hemodynamic instability. The bolus(es) should immediately be followed by a continuous infusion at 0.25-0.5 ml/kg/min. The infusion should run for a minimum of 10 minutes after the return of hemodynamic stability. However, there are documented reports of recurrent systemic toxicity even after this. For this reason, patients should be admitted for at least 12 hours for observation and additional doses of intralipid as needed for rebound symptoms or hemodynamic compromise.

Prolonged block recovery: This is not expected as the medication injected is fixed, and the drugs will be injected under ultrasound vision around nerves. If it occurs, 24 hours period will be given for observation. And if it still doesn't recover, then neurological advice will be sought.

Data collection:

This prospective study would entail the collection of the following patient-specific data:

Demographic Data: Age, gender, ASA grading, comorbidities, surgery

Lab Data: Routine blood investigations like complete blood count and coagulation profile.

Anesthesia and block details: Type of airway device, hemodynamic, block details: block name, normal/abnormal anatomy, local anaesthetics injected; rescue analgesics needed, motor assessment and complications at 30 minutes after arrival and before discharge from PACU, postoperatively in Ward at every hour till muscle power recovery and after discharge at home on day 2 and 5.

One assigned co-investigator will enter the recorded patient data with a code and no name into the password-protected master chart.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Patients undergoing AV fistula creation in the antecubital fossa

Exclusion Criteria:

* - Patient Refusal
* Hemodynamically unstable patient
* Local infection over the insertion site
* Coagulopathy
* Known allergy to Local Anaesthetic medications
* Abnormal anatomy
* Use of antiplatelet within 7 days of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Requirement of additional analgesics intraoperatively or block failure (conversion to general anaesthesia) | 20 minutes to 2 hours 30 minutes
  Paracetamol 15 mg/kg or Fentanyl 0.5 mics/kg or local infiltration or change to General Anesthesia

SECONDARY OUTCOMES:
Time of motor recovery of block | up to 24 hours
  The assessment will start from two hours after time 0 and will continue every 30 minutes till 6 hours and every hour till discharge or complete recovery of the block.
Rate of complications | up to 24 hours
  Pneumothorax, Horner syndrome, Hematoma, Diaphragmatic paralysis, Local anaesthetic systematic toxicity (LAST)

OTHER OUTCOMES:
Brachial artery diameter | 0 to 3 hours
  Brachial artery diameter will be checked before and after the block

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, MD, EDIC, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Oman

REFERENCES:
- See also: Shrestha, N. et al. (2020) "delayed neurological recovery after ultrasound-guided brachial plexus block: A case report," Local and Regional Anesthesia, Volume 13, pp. 33-35. Available at: https://doi.org/10.2147/lra.s250989 — https://doi.org/10.2147/lra.s250989
- See also: Subbiah, V. et al. (2018) "Observational study of the efficacy of supraclavicular brachial plexus block for arteriovenous fistula creation," Indian Journal of Anaesthesia, 62(8), p. 616. Available at: https://doi.org/10.4103/ija.ija_293_18. — https://doi.org/10.4103/ija.ija_293_18
- See also: Monte, A.I. et al. (2011) "Comparison between local and regional anesthesia in arteriovenous fistula creation," The Journal of Vascular Access, 12(4), pp. 331-335. Available at: https://doi.org/10.5301/jva.2011.8560. — https://pubmed.ncbi.nlm.nih.gov/21928240/
- See also: Hussien, R.M. and Ibrahim, D.A. (2018) "Ultrasound guided axillary brachial plexus block versus supraclavicular block in emergency crushed hand patients : A comparative study," The Open Anesthesia Journal, 12(1), pp. 34-41. — https://openanesthesiajournal.com/VOLUME/12/PAGE/34/FULLTEXT/
- See also: Ferré, F. et al. (2019) "Hemidiaphragmatic paralysis after ultrasound-guided supraclavicular block: A prospective cohort study," Brazilian Journal of Anesthesiology (English Edition), 69(6), pp. 580-586. — https://www.bjan-sba.org/article/doi/10.1016/j.bjane.2019.10.005
- See also: Gauss, A. et al. (2014) "Incidence of clinically symptomatic pneumothorax in ultrasound-guided infraclavicular and supraclavicular brachial plexus block," Anaesthesia, 69(4), pp. 327-336. — https://pubmed.ncbi.nlm.nih.gov/24641639/
- See also: Arab, S.A. et al. (2014) "Ultrasound-guided supraclavicular brachial plexus block," Anesthesia & Analgesia, 118(5), pp. 1120-1125. Available at: https://doi.org/10.1213/ane.0000000000000155. — https://pubmed.ncbi.nlm.nih.gov/24686046/
- See also: Bhatia, A. et al. (2010) "Pneumothorax as a complication of the ultrasound-guided supraclavicular approach for brachial plexus block," Anesthesia & Analgesia, 111(3), pp. 817-819. Available at: https://doi.org/10.1213/ane.0b013e3181e42908 — https://doi.org/10.1213/ane.0b013e3181e42908
- See also: Gao, C. et al. (2020) "Comparison of regional and local anesthesia for arteriovenous fistula creation in end-stage renal disease: A systematic review and meta-analysis." Available at: https://doi.org/10.21203/rs.3.rs-25806/v1. — https://bmcanesthesiol.biomedcentral.com/articles/10.1186/s12871-020-01136-1
- See also: Nofal, W.H. et al. (2017) "Ultrasound-guided axillary brachial plexus block versus local infiltration anesthesia for arteriovenous fistula creation at the forearm for hemodialysis in patients with chronic renal failure," Saudi Journal of Anaesthesia — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5292858/
- See also: Stav, A. et al. (2016) "Comparison of the supraclavicular, infraclavicular and axillary approaches for ultrasound-guided brachial plexus block for surgical anesthesia," Rambam Maimonides Medical Journal, 7(2) — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4839540/